CLINICAL TRIAL: NCT05644561
Title: A Phase 3, Open-label, Single-arm, Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy, Safety, and Immunogenicity of Ravulizumab Administered Intravenously in Pediatric Participants (6 to < 18 Years of Age) With Generalized Myasthenia Gravis (gMG)
Brief Title: Evaluation of Pharmacokinetics, Pharmacodynamics, Efficacy, Safety, and Immunogenicity of Ravulizumab Administered Intravenously in Pediatric Participants With Generalized Myasthenia Gravis (gMG)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-MG-319
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis; gMG
Keywords: Generalized Myasthenia Gravis; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab Intravenous (IV) Infusion (Experimental): All participants will receive a weight-based loading dose of ravulizumab IV on Day 1, followed by weight-based maintenance dose of ravulizumab on Day 15 and once every 8 weeks (q8w) thereafter for participants weighing ≥ 20 kg, or once every 4 weeks (q4w) for participants weighing < 20 kg, for a total of 122 weeks of treatment.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Ravulizumab will be administered by intravenous (IV) infusion.

SUMMARY:
The primary purpose of this study is to characterize the pharmacokinetics and pharmacodynamics of treatment with ravulizumab intravenous infusion in pediatric participants with gMG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gMG confirmed by a positive serologic test for anti-AChR antibodies (Abs) obtained at Screening and/or during Screening Period
* Myasthenia Gravis Foundation of America (MGFA) Clinical Classification of Class II to Class IV at Screening
* Participants receiving treatment must be on a stable dosing regimen of adequate duration prior to Screening and during the Screening Period.
* Eculizumab-experienced participants must have been enrolled and treated with eculizumab in Study ECU-MG-303 for at least 6 months (180 days) and must have been on a stable dose for ≥ 2 months (60 days) prior to Screening.
* All participants must be vaccinated against meningococcal infection

Exclusion Criteria:

Medical Conditions

* Any untreated thymic malignancy, carcinoma, or thymoma.
* Participants with a history of treated benign thymoma
* History of thymectomy, thymomectomy, or any thymic surgery within the 12 months prior to Screening
* History of N meningitidis infection
* Known to be human immunodeficiency virus (HIV) positive
* History of unexplained infections
* Known or suspected history of drug or alcohol abuse or dependence within 1 year prior to the start of the Screening Period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum Concentration of Ravulizumab | Day 1 predose through Week 18 predose
Serum Free C5 Concentration | Day 1 predose through Week 18 predose

SECONDARY OUTCOMES:
Change From Baseline in The Quantitative Myasthenia Gravis (QMG) Total Score at Up to Week 18 | Baseline, Up to Week 18
Change From Baseline in Myasthenia Gravis-Activities Of Daily Living (MG-ADL) Total Score at Up to Week 18 | Baseline, Up to Week 18
Change From Baseline in Myasthenia Gravis Composite (MGC) Score at Up to Week 18 | Baseline, Up to Week 18
Change in Status from Week 10 in Myasthenia Gravis Foundation of America Postintervention Status (MGFA-PIS) as Assessed by the Investigator or Neurologist at Up to Week 18 | Week 10, Up to Week 18
Change from Baseline in Neurology Quality of Life (Neuro QoL) Pediatric Fatigue Score at Up to Week 18 | Baseline, Up to Week 18
  Participants ≥8 years of age will be evaluated.
Change from Baseline in Patient-reported Outcomes Measurement Information System (PROMIS) Parent Proxy - Fatigue Score at Up to Week 18 | Baseline, Up to Week 18
  Participants <8 years of age will be evaluated.
Number of Participants With ≥5-point Reduction Compared to Baseline in the QMG Total Score Over Time Through Week 18 | Baseline through Week 18
Number of Participants With ≥3 point Reduction Compared to Baseline in the MG-ADL Total Score Over Time Through Week 18 | Baseline through Week 18
Number of Participants That Improve or Remain Stable in QMG Total Score at Week 18 Compared to Baseline | Baseline through Week 18
  Stable is defined as a ±5-point change from Baseline.
Number of Participants That Improve or Remain Stable in MG ADL Total Score at Week 18 Compared to Baseline | Baseline through Week 18
  Stable is defined as a ±3-point change from baseline.
Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events | Baseline up to Week 126 (8 weeks after last dose of study drug)
Number of Participants With Anti-Drug Antibody (ADA) at Week 18 | Baseline through Week 18

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Denton, Texas
- France (2):
  - Research Site, Marseille
  - Research Site, Paris
- Italy (3):
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Itabashi-ku, Japan
- Research Site, Leiden, Netherlands
- Research Site, Belgrade, Serbia
- Spain (2):
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR